CLINICAL TRIAL: NCT03223740
Title: A Phase III Trial of Preoperative or Postoperative Chemoradiation Therapy for Potentially Resectable Adenocarcinoma of Stomach Cancer
Brief Title: Preoperative Stomach Cancer Induction Chemotherapy and Radiation Therapy
Acronym: President
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Collaborators: Xijing Hospital (Other)
Responsible Party: Principal Investigator, ming zeng, MD, Director of Cancer Center, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: President Trial
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Locally Advanced Gastric Carcinoma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 pre-operative chemoradiation (Experimental): Chemo1 x 2 followed by ChemRT followed by Surgery followed by Chemo2 x 2
  Interventions: Other: Arm 1 pre-operative chemoradiation
- Arm 2 post operative chemoradiation (Active Comparator): Surgery followed by Chemo1 x 2 followed by ChemRT followed by Chemo2 x 2
  Interventions: Other: Arm 2 post operative chemoradiation

INTERVENTIONS:
Other: Arm 1 pre-operative chemoradiation — Chemotherapy 1:
  First 2 courses of chemotherapy with the Capacitabine /cisplatin/ combination.Capacitabine1 g/me2 day 1 to 14. Cisplatin will be given at 20 mg/m2 as a one-hour bolus on day1-5.
  Chemoradiotherapy:
  At the end of the second 21 days of chemotherapy and one week of rest (day 57), a total of 45 Gy(1.8 Gyfx/d) of radiotherapy will be given with concurrent capacitabine 625 mg/m2 and weekly Taxol 45mg/m2 over 3 hours for 5 weeks.
  Chemotherapy2:
  Four to five weeks after chemoradiotherapy, Restaged and surgical resection, a D2 resection is encouraged. Peritoneal cytology will be obtained. The J-tube will be left in for at least 8 weeks after surgery to supplement patient's nutrition.
  2nd courses of chemotherapy with the Capacitabine. Capacitabine1 g/me2 day 1 to 14. Chemotherapy will be repeated beginning on Day 29.
  Arms: Arm 1 pre-operative chemoradiation
Other: Arm 2 post operative chemoradiation — Surgical resection, a D2 resection is encouraged.
  Chemotherapy 1:
  All patients will first receive two courses of chemotherapy with the Capacitabin /cisplatin/ combination.Capacitabine1 g/me2 day 1 to 14. Cisplatin will be given at 20 mg/m2 as a bolus on day1-5. Chemotherapywill be repeated beginning on Day 22.
  Chemoradiotherapy:
  At the end of the second 21 days of chemotherapy and one week of rest (day 57), a total of 45 Gy(1.8 Gyfx/d) of radiotherapy will be given with concurrent capacitabine 625 mg/m2 and weekly Taxol 45mg/m2 over 3 hours for 5 weeks.
  Chemotherapy2:
  2nd courses of chemotherapy with the Capacitabin. Capacitabine 1g/me2 day 1 to 14. Chemotherapy will be repeated beginning on Day 29
  Arms: Arm 2 post operative chemoradiation

SUMMARY:
Based upon RTOG 9904, this study is to investigate the role of preoperative chemo and chemoradiation for locally advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with potentially resectable adenocarcinoma of the stomach with histologic proof.
* EUS or MRI stage T3-4, any N, M0.
* Adequate bone marrow (defined as peripheral absolute granulocyte count of > 2,000/μL, and platelet count of>100,000/μL), liver (bilirubin < 1.5 mg/dl), and renal functions (creatinine < 1.5 mg/dl).
* Absence of peritoneal disease by laparoscopic staging; no positive cytology of pleural, or pericardial effusion.
* No prior major surgery or radiotherapy to the stomach, or immunotherapy or chemotherapy for any reason.
* Patients must have a life expectancy of at least 16 weeks.
* Performance status of < 2 (Zubrod scale).
* No biopsy proof of lymph node metastases outside the study field.
* No evidence of metastatic disease to distant organs.
* No presence of concurrent or previous malignancies < 5 years, other than noninvasive skin cancer.
* No uncontrolled or severe cardiac disease, diabetes or hypertension.
* Signed study-specific consent form prior to study entry.

Exclusion Criteria:

* Evidence of metastatic disease
* Prior chemotherapy or radiotherapy
* Patients with a past history of cancer
* Patients with other significant underlying medical conditions that may be aggravated by the study treatment or are not controlled
* Pregnant or lactating females or female patients of childbearing potential who have not been surgically sterilized or are without adequate contraceptive measures
* Cardiac failure or Sever Pulmonary disease
* Patients with impaired gastrointestinal absorption for whatever reason
* Patients medically unfit for cisplatin or taxol chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | up to 5 year

SECONDARY OUTCOMES:
Overall Survival | up to 5 year
R0 Resection Rate | At time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zeng, MD PhD, Study Chair — Sichuan Academy of Medical Science; Hongwei Zhang, MD PhD, Study Chair — Xijing Hosptial, GI institute
Locations (3):
- China (3):
  - Xijing Hospital, GI institute, Xi’an, Shanxi
  - friendship Hospital, Chengdu, Sichuan
  - ziyang People's Hospital, Siyang, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided